CLINICAL TRIAL: NCT00184886
Title: The Influence of Methotrexate on the Metabolism and Vascular Effects of Adenosine in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MTX-Ado; ZonMw Nr. 920-03-249
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2006-02-14 (Estimated); Status verified 2006-02

CONDITIONS: Methotrexate; Vasodilation
MeSH Terms: conditions — Aneurysm | interventions — Methotrexate

INTERVENTIONS:
Drug: Methotrexate 15 mg/week for 12 weeks

SUMMARY:
In this study we aim to determine whether methotrexate influences the metabolism and vascular effects of adenosine in humans in vivo. Adenosine is an endogenous purine-nucleoside with potent anti-inflammatory effects. Also, adenosine receptor stimulation induces vasodilation, ischaemic preconditioning and many other cardiovacular effects. Previous animal studies have provided limited evidence that the anti-inflammatory effects of methotrexate are mediated by adenosine receptor stimulation. In this study, we aim to determine whether also in humans in vivo, methotretate influences endogenous adenosine. Therefore, 10 patients with inflammatory arthritis are treated with methotretxae (15 mg/week orally) for 12 weeks. Before and after treatment, vasodilation to the infusion of adenosine and dipyridamole into the brachial artery is assessed as biomarker for the endogenous adenosine concentration.

Also, blood is drawn for the determination of CRP, ESR, Adenosine deaminase activity adn homocysteine.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 year
* polyarthritis
* DAS score > 2.5

Exclusion Criteria:

* previous use of MTX
* concomitant use of dipyridamole/sulfazalasine
* Alcohol > 21 U/week
* elevated liver enzymes
* pregnancy, breast-feeding, asthma, renal insufficiency, thrombocytopenia, leucocytopenia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2003-11; Study Completion 2005-01

PRIMARY OUTCOMES:
Vasodilator response to infusion of adenosine and dipyridamole into the brachial artery

SECONDARY OUTCOMES:
Adenosine deaminase activity
CRP, BSE, DAS

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Rongen, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands